CLINICAL TRIAL: NCT04040764
Title: The Tritanium Uncemented Prosthesis Versus the Cemented Triathlon Prosthesis
Brief Title: Uncemented Tritanium TKR vs Cemented Triathlon TKR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003957
Record Dates: First submitted 2019-07-12; First posted 2019-08-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: An internal pilot study comparing 2 different types of knee prosthesis; uncemented vs cemented total knee replacement
Who Masked: Participant, Outcomes Assessor
Masking Description: The following people will be blinded as to which arm of the study the patient is allocated to:
  * The patient
  * The statistician who performs the analysis of the results
  * The radiographer reporting upon the DXA scan results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uncemented Tritanium Knee Replacement (Experimental): 30 participants will be randomly allocated to receive an uncemented Tritanium total knee replacement.
  Interventions: Procedure: Tritanium uncemented Total Knee Replacement
- Cemented Triathlon Knee Replacement (Active Comparator): 30 participants will be randomly allocated to receive standard Triathlon cemented total knee replacements.
  Interventions: Procedure: Tritanium uncemented Total Knee Replacement

INTERVENTIONS:
Procedure: Tritanium uncemented Total Knee Replacement — This will be an internal pilot study in which patients will be blinded and randomly assigned to 1 of 2 arms with 30 patients in each arm. The first arm will receive a Triathlon knee replacement device which is cemented into place. The second arm will receive an uncemented Triathlon Tritanium TKR.
  Other Names: Triathlon Cemented Total Knee Replacement

SUMMARY:
The Study aims to investigate whether there is a clinically important difference in peri-articular bone mineral density (BMD) and trabecular bone score (TBS) between patients undergoing two different types of knee replacement fixation - uncemented Tritanium total knee replacement (TKR) and cemented Triathlon TKR.

Before undertaking a full randomised control trial however, it is necessary to establish that the proposed methodology and approach are feasible. Therefore an internal pilot study will be performed first. This registration is for the internal pilot study.

DETAILED DESCRIPTION:
There have been many studies published that have shown a reduction in bone density around knee replacements. Exact reasons for this are not fully understood but one theory is that the stresses transmitted to the bone around a new knee replacement do not adequately load the surrounding bone due to the stress shielding effects of the cement. Bone requires itself to be loaded by weight-bearing pressure in order to maintain its density and structural integrity.

A loss of bone density around the knee has potentially significant consequences for patients. The ability of the bone to support the knee replacement may be compromised, potentially leading to subsidence and failure of the joint replacement. Patients are known to be more prone to falls within 1 year of having a TKR in comparison to age matched controls who have not undergone knee replacements. The incidence of falls following knee replacement was shown to be 38% in one study after the first year post-operatively, compared to 24% in non-TKR subjects. A reduction in bone density following TKR also renders patients more prone to aseptic loosening and fracture around the knee replacement with potentially disastrous consequences.

The majority of research seems to demonstrate a loss of BMD around the knee at around 12 months following TKR surgery, with the most significant BMD decrease occurring between the period of 5-12 weeks post-surgery, occurring primarily at the periprosthetic region. Up to 68% of patients have been reported as showing BMD loss after TKR at the distal anterior femur within the first 12 months post-operatively. The possible fracture risk associated with this has been investigated. Women aged ≥ 70 years who have undergone TKR surgery are 1.6 times more likely to have a fracture than younger patients and 2.3 times more likely to suffer a fracture than men.

Bone density is measured by use of Dual X-ray Absorbitometry scans (DEXA). However, DEXA bone density measurement alone provides an incomplete picture of bone strength. DEXA measurement is derived from the bone mineral content (BMC) divided by bone area, but does not account for the distribution of the trabeculae and the structural integrity of the microarchitecture. This has led to the development of a tool called the trabecular bone score (TBS) which is able to differentiate between microarchitectures that exhibit the same density.

Advancement in technology has led to re-designs in uncemented knee replacements. These newer implants are able to withstand torsional stresses that previously would have concerned surgeons who feared implant movement in the early post-operative phase. The development of biologic coatings on to TKR components also means that bony on-growth and thus stability of the knee implant is achieved much more quickly than was previously. Surgeons have become keener to use such uncemented devices and recent research has shown comparable results in terms of patient satisfaction, Oxford Knee Scores and the need for revision surgery between cemented and uncemented devices.

Bone architecture responds to the stresses placed upon it. Theoretically, cementless fixation could help preserve periprosthetic bone stock. In uncemented total knee replacements' weight-bearing loads are transmitted through the prosthesis directly to the surrounding bone as opposed to being dissipated by a layer of cement between the implant and the periprosthetic bone. Other potential benefits of cementless fixation include shorter operating room time, ease of revision, and the elimination of complications associated with cemented fixation, including debridement of the cement and resulting loose fragments. Patterns of wear (osteolysis) can occur in cemented implants, it is hoped that the new generation of highly porous uncemented implants will enable biological bony fixation of the implant, thus providing greater osseous integration and more durable fixation.

If the number of TKR continues to rise as predicted, the economic consequences for the NHS are significant. Further clarity on the potential benefits of one implant over another is required to contribute to our knowledge of best practice and evaluate cost effectiveness.

The Triathlon cemented knee replacement has been used worldwide since 2004. A new version of the implant has been developed, this newer version has the same geometry as the Triathlon TKR but has been designed with a special biological coating which enables it to be used without cement, it is currently in use in the US. We would like to assess the potential of this implant to reduce bone density loss around the knee and to see if this will reduce the risk of bone fracture. At the same time we would like to ensure at least the non-inferiority of the uncemented implant compared to the cemented one both in terms of patient satisfaction, functional ability and improvement. We would also like to evaluate cost effectiveness of the two methods of fixation; to see if the shorter operating time associated with not using cement will result in significant cost saving for the NHS.

Before undertaking a full randomised control trial investigating the above, we would like to establish that the proposed methodology and approach are feasible. Therefore an internal pilot study will be performed first.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary TKR at the RD+E Hospital
* Patients must have completed a consent form for the study
* Patients must be prepared to comply with the pre and post-operative investigations, attendance schedule and questionnaire schedule of the study
* If the knee for surgery is suitable for standard condylar TKR components
* The diagnosis is of tricompartmental osteoarthritis of the knee
* Aged 50-70 years at time of surgery

Exclusion Criteria:

* Refusal to consent to the study
* If the knee for surgery is not suitable for standard condylar TKR.
* Pregnancy
* Prisoners
* A patient known to have substance abuse or psychological disorders that could interfere with their ability to comply with the assessment schedules
* Patients unable to read or understand the patient information leaflet and consent form
* Patients who have a Body Mass Index (BMI) ≥ 38
* Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation
* Patient has received any orthopaedic surgical intervention to the lower extremities within the past year or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the TKR to be enrolled in this study, within the next year
* Patient requires bilateral total knee replacements, or has a history of unsuccessful contralateral partial or total knee replacement
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days)
* Patients currently taking bisphosphonate medication or have taken within the previous 10 years
* The presence of peri-articular cysts evident on the pre-operative x-ray such as could compromise the stability at the bone implant interface if the uncemented component is used
* A past history of tibial or femoral osteotomy surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assessment and comparison of Trabecular Bone Score (TBS) between patients undergoing two different types of knee replacement fixation - uncemented Tritanium knee replacement and cemented Triathlon knee replacement. | Our primary outcome is TBS scores at 12 months post total knee replacement
  We plan to compareTBS data between patients randomised to the 2 arms of the trial: the uncemented Tritanium and cemented Triathlon total knee replacement. TBS is a texture parameter that evaluates gray-level pixel-by-pixel variations and provides an assessment of fracture risk. TBS is calculated from patients DEXA scan results and is in a numerical format. Baseline TBS scores will be calculated from pre-operative DEXA scans and will be compared to post op scores. Any differences in TBS scores will be compared between participants in the 2 arms of the trial.

SECONDARY OUTCOMES:
Assessment and comparison of Trabecular Bone Score (TBS) between patients undergoing two different types of knee replacement fixation - Uncemented Tritanium knee replacement and cemented Triathlon knee replacement. | 6 weeks and 6 months post-op.
  We plan to compareTBS data between patients randomised to the 2 arms of the trial: the uncemented Tritanium and cemented Triathlon total knee replacement. TBS is a texture parameter that evaluates gray-level pixel-by-pixel variations and provides an assessment of fracture risk. TBS is calculated from patients DEXA scan results and is in a numerical format. Baseline TBS scores will be calculated from pre-operative DEXA scans and will be compared to post op scores. Any differences in TBS scores will be compared between participants in the 2 arms of the trial.
Oxford Knee Score: Patient reported outcome measure (PROM) | Pre-operatively, 6 weeks post op, 6 and 12 months post op.
  The Oxford Knee Score (OKS) is a Patient Reported Outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty. The OKS consists of twelve questions covering function and pain associated with the knee. It has a scoring range of between 0-48 with the lowest score indicating the worst possible outcome and the highest score the best.
The Forgotten Joint Score (FJS): Patient reported outcome measure (PROM) | Pre-operatively, 6 weeks post op, 6 and 12 months post op.
  The FJS will focus on the patients' awareness of their joint replacement during a range of day to day and recreational activities. It is a validated PROM and consists of 12 questions where subjects are asked to rate their awareness of their joint replacement during various activities. The range of scoring is from 0-100, high scores indicate good outcome, that is, a high degree of forgetting the joint.
The Knee Injury and Osteoarthritis Outcome Score (KOOS): Patient reported outcome measure (PROM) | Pre-operatively, 6 weeks post op, 6 and 12 months post op.
  The KOOS questionnaire is designed to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardised answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
EQ5D: Patient reported outcome measure (PROM) | Pre-operatively, 6 weeks post op, 6 and 12 months post op.
  The EQ5D PROM will be used as a measure of health-related quality of life. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This will be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Hospital Anxiety and Depression Scale (HADS): Patient reported outcome measure (PROM) | Pre-operatively, 6 weeks post op, 6 and 12 months post op.
  The HADS PROM will be used to determine levels of anxiety and depression in participants. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression with higher numbers depicting higher levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Waterson, MD, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust Hospital
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As this is an internal pilot study it is hoped that the data collected from this trial confirms that the methodology and approach are feasible and allows us to progress to a larger randomised control trial.

REFERENCES:
- [Background] Fricka KB, Sritulanondha S, McAsey CJ. To Cement or Not? Two-Year Results of a Prospective, Randomized Study Comparing Cemented Vs. Cementless Total Knee Arthroplasty (TKA). J Arthroplasty. 2015 Sep;30(9 Suppl):55-8. doi: 10.1016/j.arth.2015.04.049. Epub 2015 Jun 3. PMID 26118567
- [Background] Gundry M, Hopkins S, Knapp K. A Review on Bone Mineral Density Loss in Total Knee Replacements Leading to Increased Fracture Risk. Clin Rev Bone Miner Metab. 2017;15(4):162-174. doi: 10.1007/s12018-017-9238-4. Epub 2017 Oct 27. PMID 29213219
- [Background] Minoda Y, Kobayashi A, Ikebuchi M, Iwaki H, Inori F, Nakamura H. Porous tantalum tibial component prevents periprosthetic loss of bone mineral density after total knee arthroplasty for five years-a matched cohort study. J Arthroplasty. 2013 Dec;28(10):1760-4. doi: 10.1016/j.arth.2013.03.031. Epub 2013 Apr 30. PMID 23642446
- [Background] Winther N, Jensen C, Petersen M, Lind T, Schroder H, Petersen M. Changes in bone mineral density of the proximal tibia after uncemented total knee arthroplasty. A prospective randomized study. Int Orthop. 2016 Feb;40(2):285-94. doi: 10.1007/s00264-015-2852-1. Epub 2015 Jul 17. PMID 26183139
- [Background] Abu-Rajab RB, Watson WS, Walker B, Roberts J, Gallacher SJ, Meek RM. Peri-prosthetic bone mineral density after total knee arthroplasty. Cemented versus cementless fixation. J Bone Joint Surg Br. 2006 May;88(5):606-13. doi: 10.1302/0301-620X.88B5.16893. PMID 16645105
- [Background] Nam D, Kopinski JE, Meyer Z, Rames RD, Nunley RM, Barrack RL. Perioperative and Early Postoperative Comparison of a Modern Cemented and Cementless Total Knee Arthroplasty of the Same Design. J Arthroplasty. 2017 Jul;32(7):2151-2155. doi: 10.1016/j.arth.2017.01.051. Epub 2017 Feb 7. PMID 28238584